CLINICAL TRIAL: NCT01704612
Title: Comparison of Subgluteal Sciatic Nerve Block Duration in Type-2 Diabetic and Non Diabetic Patients
Brief Title: Evaluation of Block Duration in Type 2 Diabetes Patients
Acronym: Diabeteblock
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pierre and Marie Curie University (Other)
Collaborators: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Principal Investigator, Philippe Cuvillon, MD, PhD, Centre Hospitalier Universitaire de Nīmes
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-PC001
Record Dates: First submitted 2012-10-07; First posted 2012-10-11 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Diabetes Type 2
Keywords: local anesthetic; sciatic; diabetes; block; duration
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Bites and Stings | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diabete group (Active Comparator): Patient with type 2 diabete received 20 mL ropivacaine
  Interventions: Drug: ropivacaine
- Control group (Sham Comparator): no diabete reveived 20 mL ropivacaine
  Interventions: Drug: ropivacaine

INTERVENTIONS:
Drug: ropivacaine — patients received 20 mL ropivacaine 5 mg/mL on subgluteal nerve
  Other Names: naropin

SUMMARY:
Diabete animal studies demonstrated a longer period recovery after local anesthetic injection (perineural administration). No clinical study demonstrated a prolonged nerve block duration in diabete type 2 patients after peripheral nerve block. The investigators hypothesized that block recovery is delayed in diabetic patients.

DETAILED DESCRIPTION:
For diabetic patients, peripheral nerve block is an interesting alternative to general anesthesia because it provides effective analgesia and may decrease haemodynamic complication. The fear of nerve injury after regional anaesthesia in diabetic patients is a concern that has neither been confirmed nor refuted by current literature. As a matter of fact, diabetic patients with neuropathy may be considered at increased risk because of the possibility for double crush syndrome when a chronic axon lesion related to diabetes is associated with an unexpected distal nerve injury related to regional anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* age (50 80 yrs) with monofilament test 10 g (> 4/8)

Exclusion Criteria:

* refusal of sciatic nerve block,
* age < 50 yr or > 80 yr,
* American Society of Anesthesiologists state > IV,
* presence of contraindications to local anaesthesia (known allergy to local anaesthetics, sepsis),
* emergency surgery,
* patients unlikely to be fully cooperative during the study,
* psychiatric disorders, or
* those abusing alcohol or drugs, and
* participation in another study within the previous 30 days. Moreover, patients with preoperative estimated values of creatinine clearance < 50 mL min-1 (Cockroft and Gault Formula) or with glycosylated hemoglobin (A1c) level > 8 % or with type 1 diabetes mellitus (insulin therapy)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
the duration of sensory block in hours | Day 0
  The beginning of this term is defined by the end of the sciatic block injection, and the end of this period is defined by the reappearance of sensitivity to pin-prick test

SECONDARY OUTCOMES:
the duration of motor sciatic block | Day 0
  The beginning of this term is defined by the end of the sciatic block injection, and the end of this period is defined by the reappearance of motor function

OTHER OUTCOMES:
Time necessary for onset sensory and motor block time in minutes | Day 0
  peroperative period
Failure of the block: yes/no | Day 0
  perop
occurrence of neurological omplications, yes/no | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Cuvillon, PhD, Principal Investigator — APHP Pitié Salpetriere
Locations (1):
- APHP Pitié-Sampetriere, Paris, France

REFERENCES:
- [Derived] Cuvillon P, Reubrecht V, Zoric L, Lemoine L, Belin M, Ducombs O, Birenbaum A, Riou B, Langeron O. Comparison of subgluteal sciatic nerve block duration in type 2 diabetic and non-diabetic patients. Br J Anaesth. 2013 May;110(5):823-30. doi: 10.1093/bja/aes496. Epub 2013 Jan 24. PMID 23348203